CLINICAL TRIAL: NCT06852586
Title: Comparison of Postoperative Sensitivity in Posterior Teeth Using Conventional and Bulkfill Composites
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: 28 Military Dental Centre Lahore (Other Government)
Responsible Party: Principal Investigator, Zahra Zubair, Dr Zahra Zubair, 28 Military Dental Centre Lahore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: COMPOSITES
Record Dates: First submitted 2025-02-25; First posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2022-06

CONDITIONS: Class I Dental Caries
Keywords: Conventional nanohybrid composites, Bulk fill composites

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Conventional Nano-hybrid composites (Experimental): Coltene Brilliant NG Conventional Nanohybrid composites
  Interventions: Device: conventional nanohybrid composites
- Bulk fill composites (Experimental): Coltene Fillup! Bulk fill COMPOSITES
  Interventions: Device: Bulk fill composites

INTERVENTIONS:
Device: conventional nanohybrid composites — Incremental layering technique is used for restoration
  Other Names: Coltene Brilliant NG conventional Nanohybrid
  Arms: Conventional Nano-hybrid composites
Device: Bulk fill composites — Single increment in bulk form is applied for restoration
  Other Names: Coltene Fill up! BULKFILL
  Arms: Bulk fill composites

SUMMARY:
The purpose of this study is to compare the onset and severity of pain and postoperative sensitivity in patients after using conventional nanohybrid and bulkfill composites

Null Hypothesis:

There is no significant difference in mean postoperative sensitivity exhibited with conventional nano-hybrid versus bulkfill composites in mandibular molars with class 1 cavity.

DETAILED DESCRIPTION:
The study will include 79 patients with class 1 carious mandibular molars. Teeth are divided into two groups based on composite placement techniques. In group 1, 39 patients are restored with conventional nanohybrid composites using an incremental layering technique. In group 2, 40 patients are restored with bulk-fill composites containing a single increment. After taking a brief history, informed consent will be taken from patients. The depth of the cavity will be determined using a periodontal probe not extending more than 3 mm. Preoperatively, pulp vitality will be assessed using the cold thermal test. A preoperative radiograph will also be taken. A rubber dam will be used. The cavity will be prepared and a selective etch technique will be used. Patients will be recalled after 24 hours and 1 week, thermal cold tests will be performed and a questionnaire containing the Numerical Rating Scale will be given to each patient for evaluation of post-operative pain felt after 24 hours and 1 week.

ELIGIBILITY:
Inclusion Criteria:

- 1. Patients with ages range from 18- 55 years. 2. Male/ Female. 3. Mandibular molars with class 1 shallow-sized cavity with no history of pre-operative pain or sensitivity.

4. Ability to understand the use of pain and sensitivity scale. 5. Patients with adequate oral hygiene and willingness to participate in this study.

Exclusion Criteria:

- 1. Patients with deep caries of tooth associated with pain and sensitivity. 2. Patients who have consumed any type of medication before treatment. 3. Periapical pathologies (periapical abscess, sinus tract, periapical cyst, pulpal abscess.

4. Unfavorable location of the tooth, severe tooth malposition, and trismus.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 79 (Actual)
Dates: Start 2022-08-26 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Avoidance of Postoperative sensitivity in posterior class 1 carious mandibular molars restored with composites | 24 hours and 1 week after restoring Class 1 caries
  Numerical Rating Scale

CONTACTS AND LOCATIONS:
Overall Officials: Zahra Zubair, BDS, Principal Investigator — 28 Military Dental Centre
Locations (1):
- Zahra Zubir, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Name, Gender, Age, and Tooth no., Diagnosed class 1 caries
Time Frame: 6 months after publication
Access Criteria: zahra_zubair@hotmail.com

REFERENCES:
- [Background] Afifi SMH, Haridy MF, Farid MR. Evaluation of Post-Operative Sensitivity of Bulk Fill Resin Composite versus Nano Resin Composite: A Randomized Controlled Clinical Study. Open Access Maced J Med Sci. 2019 Jul 26;7(14):2335-2342. doi: 10.3889/oamjms.2019.656. eCollection 2019 Jul 30. PMID 31592052
- [Background] Cieplik F, Scholz KJ, Anthony JC, Tabenski I, Ettenberger S, Hiller KA, Buchalla W, Federlin M. One-year results of a novel self-adhesive bulk-fill restorative and a conventional bulk-fill composite in class II cavities-a randomized clinical split-mouth study. Clin Oral Investig. 2022 Jan;26(1):449-461. doi: 10.1007/s00784-021-04019-y. Epub 2021 Jun 15. PMID 34129074
- [Background] Tardem C, Albuquerque EG, Lopes LS, Marins SS, Calazans FS, Poubel LA, Barcelos R, Barceleiro MO. Clinical time and postoperative sensitivity after use of bulk-fill (syringe and capsule) vs. incremental filling composites: a randomized clinical trial. Braz Oral Res. 2019 Sep 16;33(0):e089. doi: 10.1590/1807-3107bor-2019.vol33.0089. PMID 31531552
- [Background] Chiodera G, Orsini G, Tosco V, Monterubbianesi R, Manauta J, Devoto W, Putignano A. Essential Lines: a simplified filling and modeling technique for direct posterior composite restorations. Int J Esthet Dent. 2021 May 10;16(2):168-184. PMID 33969973
- [Background] Veloso SRM, Lemos CAA, de Moraes SLD, do Egito Vasconcelos BC, Pellizzer EP, de Melo Monteiro GQ. Clinical performance of bulk-fill and conventional resin composite restorations in posterior teeth: a systematic review and meta-analysis. Clin Oral Investig. 2019 Jan;23(1):221-233. doi: 10.1007/s00784-018-2429-7. Epub 2018 Mar 28. PMID 29594349
- [Background] Nascimento AS, Rodrigues JFB, Torres RHN, Santos KO, Fook MVL, Albuquerque MS, Lima EA, Filgueira PTD, Santos JBMD, Oliveira LJR, Braz R. Physicomechanical and thermal analysis of bulk-fill and conventional composites. Braz Oral Res. 2019 Mar 18;33:e008. doi: 10.1590/1807-3107bor-2019.vol33.0008. PMID 30892408
- [Background] Yazici AR, Kutuk ZB, Ergin E, Karahan S, Antonson SA. Six-year clinical evaluation of bulk-fill and nanofill resin composite restorations. Clin Oral Investig. 2022 Jan;26(1):417-426. doi: 10.1007/s00784-021-04015-2. Epub 2021 Jun 10. PMID 34110494
- [Background] Burke FJT, Mackenzie L. Bonding to dentine: an update on universal adhesives. Dent Update. 2021;48(8):620-31. doi: 10.12968/denu.2021.48.8.620.
- [Background] Burke FJT, Mackenzie L, Sands P, Shortall ACC. Ten tips for avoiding post-operative sensitivity with posterior composite restorations. Dent Update. 2021;48(10):823-32. DOI: 10.12968/denu.2021.48.10.823.